CLINICAL TRIAL: NCT07296185
Title: The Effect of Body Awareness on Pain, Disability, Sensorimotor Acuity, Psychosocial and Central Sensitization Levels in Individuals With Non-Specific Chronic Low Back Pain
Status: Not yet recruiting | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Rabia Ece KESKİN, Principal Investigator, Physiotherapist, Medipol University
Other Study IDs: KBA-MED25-REK; E-10840098-202.3.02-624 (Other: Istanbul Medipol University Ethics Committee)
Record Dates: First submitted 2025-07-03; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Non-specific Chronic Low Back Pain
Keywords: Body awareness; Central sensitization; Sensorimotor Acuity; Disability; Non-specific Chronic Low Back Pain; Psychosocial Factor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-specific Chronic Low Back Pain Group (NCLBP Group): A total of forty-one individuals with non-specific chronic low back pain will be included in the NCLBP group (n=41). All participants will be between 25 and 65 years of age. Pain levels and catastrophization levels of the patients with NCLBP individuals will be assessed using the Visual Analogue Scale (VAS) and Pain Catastrophizing Scale (PCS). Lumbar joint position sense will be evaluted using a with digital electrogoniometer, tactile acuity of the lumbar region will be assessed using Two-Point Discrimination Test (TPDT), Pressure Pain Threshold (PPT) will be measured using algometer, functionality will be assessed using Roland Morris Disability Questionnaire (RMDQ), body awareness levels with Fremantle Back Awareness Questionnaire (FreBAQ) and central sensitization levels with Central Sensitization Inventory (CSI).
  Interventions: Other: No intervention
- Healthy Controls (Healthy Group): A total of forty-one healthy individuals will be included in the healthy group (n=41). All participants will be between 25 and 65 years of age. Pain levels and catastrophization levels of the healthy individuals will be assessed using the Visual Analogue Scale (VAS) and Pain Catastrophizing Scale (PCS). Lumbar joint position sense will be evaluted using a with digital electrogoniometer, tactile acuity of the lumbar region will be assessed using Two-Point Discrimination Test (TPDT), Pressure Pain Threshold (PPT) will be measured using algometer, functionality will be assessed using Roland Morris Disability Questionnaire (RMDQ), body awareness levels with Fremantle Back Awareness Questionnaire (FreBAQ) and central sensitization levels with Central Sensitization Inventory (CSI).
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention applied, observational study.

SUMMARY:
This study will be conducted to examine the levels of pain, pressure pain threshold, joint position sense, sensation, functionality, pain catastrophizing, central sensitization, and body awareness in individuals with non-specific chronic low back pain, and to compare these findings with those of healthy individuals. Additionally, the study will aim to objectively investigate the relationships between lumbar self-perception (FreBAQ) and tactile acuity (TPDT), pressure pain threshold (PPT), lumbar joint position sense (LJPS), as well as psychosocial (PCS) and central sensitization (CSI) indicators in individuals with non-specific chronic low back pain. Furthermore, the study will seek to evaluate the predictive effects of lumbar self-perception on pain (VAS) and disability (RMDQ), in conjunction with objectively assessed sensory and sensorimotor measures in individuals with non-specific chronic low back pain.

DETAILED DESCRIPTION:
This study will be conducted to examine the levels of pain, pressure pain threshold, joint position sense, sensation, functionality, pain catastrophizing, central sensitization, and body awareness in individuals with non-specific chronic low back pain, and to compare these findings with those of healthy individuals. Additionally, the study will aim to objectively investigate the relationships between lumbar self-perception (FreBAQ) and tactile acuity (TPDT), pressure pain threshold (PPT), lumbar joint position sense (LJPS), as well as psychosocial (PCS) and central sensitization (CSI) indicators in individuals with non-specific chronic low back pain. Furthermore, the study will seek to evaluate the predictive effects of lumbar self-perception on pain (VAS) and disability (RMDQ), in conjunction with objectively assessed sensory and sensorimotor measures in individuals with non-specific chronic low back pain. A total of forty-one individuals with non-specific chronic low back pain will be included in the NCLBP group (n=41), and forty-one healthy individuals will be included in the healthy group (n=41). All participants will be between 25 and 65 years of age. Pain levels and catastrophization levels of all participants will be assessed using the Visual Analogue Scale (VAS) and Pain Catastrophizing Scale (PCS). Lumbar joint position sense will be evaluted using a with digital electrogoniometer, tactile acuity of the lumbar region will be assessed using Two-Point Discrimination Test (TPDT), Pressure Pain Threshold (PPT) will be measured using algometer, functionality will be assessed using Roland Morris Disability Questionnaire (RMDQ), body awareness levels with Fremantle Back Awareness Questionnaire (FreBAQ) and central sensitization levels with Central Sensitization Inventory (CSI).

ELIGIBILITY:
Inclusion criteria are as follows:

* Eligible participants were defined according to the National Institute of Health Task Force for Research Standards for Chronic Pain (RTF). The RTF defines chronic pain as a pain problem that has persisted for at least 3 months and has been present on at least half of the days in the past 6 months. Following these guidelines, two questions will be used to determine chronicity:

  1. "How long has the pain been an ongoing problem for you?"
  2. "How often has pain been an ongoing problem for you over the past 6 months?" A response of "greater than 3 months" to question 1 and "at least half the days in the past 6 months" to question 2 indicated chronic pain.
* Being 25 and 65 years of age and having no spinal fractures or acute disc herniation;
* Non-specific chronic low back group for pain a current VAS pain rating ≥4/10; and scoring at least 4 points on the Roland-Morris Disability Questionnaire (RMDQ),
* Having pain that does not correspond to specific anatomical structures and is widespread;
* Having no current psychiatric disorders or cognitive impairments and cognitive level sufficient to complete the interview and questionnaires;
* For the healthy group; Absence of low back pain during the past six months, no history of chronic pain lasting ≥3 months in any body region, having a Visual Analog Scale (VAS) score of VAS ≤1, which having a Roland Morris Disability Questionnaire (RMDQ) score of RMDQ ≤4;
* Having no history of spinal surgery.

Exclusion criteria are as follows:

* The current use of tranquilizers or opioids, any visual or motor impairments (including dyslexia) or presentation with any neurological disease or significant mental illness;
* Potential subjects if they have nerve symptoms below the knee;
* Diagnosed chronic fatigue syndrome, fibromyalgia, or other chronic widespread pain syndromes.
* Severe comorbidities such as neurological disorders, cardiovascular diseases, or rheumatologic conditions.
* Patients who had undergone spinal surgery, had any illness, or received any treatment that could cause harm were excluded;
* Having a diagnosis of lumbar radiculopathy;
* Tumors or infections;
* Pain arising from metastasis, osteoporosis, inflammatory arthritis, or fractures;
* Specific medical conditions (such as neck or back surgery within the last 3 years, osteoporotic vertebral fractures);
* Receiving any other treatment for chronic non-specific low back pain during the study period.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of forty-one individuals with non-specific chronic low back pain will be included in the NCLBP group (n = 41), and forty-one healthy individuals will be included in the healthy group (n = 41). All participants will be between 25 and 65 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Central sensitization levels | Baseline.
  Central Sensitization levels will be assessed using the Central Sensitization Inventory (CSI). The CSI consists of 25 items that evaluate somatic and emotional health-related symptoms commonly observed in conditions associated with central sensitization. Each item is rated on a 5-point temporal Likert scale with the following numerical options: Never (0), Rarely (1), Sometimes (2), Often (3), and Always (4). The total score ranges from 0 to 100. Higher scores indicate greater symptom severity (15).
Body awareness levels | Baseline.
  Body awareness level will be assessed using the Fremantle Back Awareness Questionnaire (FBAQ). The FBAQ is a questionnaire that assesses body awareness related to the low back. The questionnaire consists of nine questions. Each item is scored from 0 to 4. The FBFQ total score ranges from 0 to 36. Higher scores indicate greater disruption in low back-specific body awareness.
Tactile acuity of the lumbar region | Baseline.
  Tactile acuity of the lumbar region will be assessed using the Two-Point Discrimination Test (TPDT) with a mechanical esthesiometer. The TPDT consists of three ascending and three descending series for the right and left sides. The TPDT score is calculated as the average of three ascending and three descending thresholds for each side. The right and left TPTD values are then averaged, and the left ascending and left descending values are then averaged. The right and left TPDT values are then averaged to obtain a total TPDT score representing the overall tactile acuity of the lumbar spine.Lower values indicate better tactile acuity.
Lumbar joint position sense | Baseline.
  Lumbar joint position sense (LJPS) will be measured using with digital electrogoniometer. LJPS errors will be recorded in degrees during lumbar flexion, extension, and left and right lateral flexion movements, and these values will be used as an estimate of lumbar proprioceptive accuracy. Each test will be repeated three times, and the average of the three trials was used for analysis. Repositioning errors will be calculated as the difference between the actual angle and the target angle in degrees.Greater absolute repositioning errors demonstrate poorer lumbar position sense.
Pressure Pain Threshold (PPT) | Baseline.
  Pressure pain thresholds (i.e., the minimum pressure point that causes an unpleasant sensation) will be measured using a handheld pressure algometer with a 1 cm2 circular probe surface that allows measurement of pressure force up to 10 kg (Baseline®, 22 lbs × 1⁄4 lb and 10 kg ×). The measurement points will be bilaterally, 2 cm lateral to the L5 spinous process and the plantar side of the second toe. Three measurements will be taken at 30-second intervals for each area, and the average of these three measurements will be used for data analysis. Higher algometer values indicate an increased pressure pain threshold. Data will be recorded in kg/cm².
Pain levels | Baseline.
  Participants pain levels will be measured using Visual Analog Scale (VAS). Participants will be asked to rate the intensity of pain they have experienced over the past week. A 10-cm continuous line will be presented, with one end labeled 'No pain at all' and the other end labeled 'Unbearable pain.' Participants will be asked to mark the level of their pain intensity on a 10-cm horizontal line with '0' at the beginning and '10' at the end. The marked location will then be measured using a ruler and recorded in centimeters. On the Visual Analog Scale (VAS), higher scores indicate greater pain intensity.
Functionality | Baseline.
  The Roland Morris Disability Questionnaire (RMDQ) will be used to measure participants functional limitations. The RMDQ is a 24-item questionnaire that assesses normal activities of daily living. Participants will be asked to mark the items they found difficult to perform due to their chronic low back pain. Each response is scored as "no" (difficulty = 0 points) or "yes" (difficulty = 1 point). Total scores range from 0 to 24, with higher scores indicating more severe disability.
Catastrophization levels | Baseline.
  The Pain Catastrophizing Scale (PCS) will be used to assess the catastrophizing levels of the participants. The PCS consists of 13 items that measure catastrophic thinking and maladaptive responses to pain, and includes three subscales assessing helplessness, magnification, and rumination. For each item, participants will be asked to choose one of the following options: none = 0, mild = 1, moderate = 2, considerable = 3, or always = 4. The PCS total score ranges from 0 to 52, with higher scores indicating more destructive thoughts and feelings related to pain.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar KAYA SARIBAŞ, PhD, Study Chair — Medipol University
Locations (1):
- Istanbul Medipol Unıversity, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No